INFORMED CONSENT VERSION: 1 DATE: 28<sup>TH</sup> JUNE 2019

## CONSENT BY PATIENT FOR CLINICAL RESEARCH

| I,(Name of Patient) Identity Card No |
|---|
| of |
| (Address) |
| hereby agree to take part in the clinical research (clinical study/questionnaire study/drug trial) specified below: |
| <u>Title of Study:</u> The Effects of Platelet-Rich Plasma vs Prolotherapy Injection on Functional and Pain Scores in Supraspinatus Tendinopathy: A Randomized Controlled Trial. |
| the nature and purpose of which has been explained to me by: |
| Dr: |
| Sports Medicine Specialist |
| and interpreted by(Name & Designation of Interpreter) |
| to the best of his/her ability in English language/dialect. |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. |
| Date: Signature or Thumbprint |
| (Patient) |
| IN THE PRESENCE OF |

INFORMED CONSENT VERSION: 1 DATE: 28<sup>TH</sup> JUNE 2019

| Name) | |
|---|---|
| ) Identity Card No) Signature | |
| (Witness for Signature of Patient) | |
| Designation) | |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. | |
| Date Signature | |
| (Attending Doctor) | |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research Date | • |

CONSENT BY PATIENT FOR

(Attach patient's sticker here)